CLINICAL TRIAL: NCT01883596
Title: Chlorhexidine Gluconate for Prevention of Ventilator Associated Pneumonia in a Pediatric Intensive Care Unit.
Brief Title: Chlorhexidine Gluconate for Prevention of Ventilator Associated Pneumonia in Children.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sinaloa Pediatric Hospital (Other)
Responsible Party: Principal Investigator, Jesús Javier Martínez-García, MD, Sinaloa Pediatric Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HPS-02
Record Dates: First submitted 2013-06-11; First posted 2013-06-21 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Mechanical Ventilation for More Than 48 Hours.
MeSH Terms: interventions — chlorhexidine gluconate; Chlorhexidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 0.12% Chlorhexidine (Experimental): Bexident® (0.12% chlorhexidine) solution, applied topically, every 8 hrs.
  Interventions: Drug: 0.12% chlorhexidine solution
- Placebo (Placebo Comparator): 7.4% alcohol, glycerine, normal saline solution, applied topically, every 8 hrs.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 0.12% chlorhexidine solution — Bexident® (0.12% chlorhexidine solution)
  Other Names: Peridex, Betasept, PerioGard.
  Arms: 0.12% Chlorhexidine
Drug: Placebo — 7.4% alcohol, glycerine, normal saline solution, applied topically, every 8 hrs.
  Arms: Placebo

SUMMARY:
To determine the efficacy of prophylaxis with 0.12% chlorhexidine gluconate compared with placebo to prevent ventilator associated pneumonia in children admitted to a pediatric critical care unit.

DETAILED DESCRIPTION:
Randomised controlled trial to determine the efficacy of 0.12% chlorhexidine gluconate compared with placebo to prevent ventilator associated pneumonia in children admitted to a pediatric critical care unit.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1 month to 18 years admitted to the intensive care unit.
* Intubated for more than 48 hours.

Exclusion Criteria:

* Clinical or radiological diagnosis of pneumonia previous to the endotracheal intubation.
* Allergy to chlorhexidine.
* Known immune deficiency.

Elimination Criteria:

* Transfer to another hospital.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2012-10; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of ventilator associated pneumonia | Participants will be followed for the duration of intensive care unit stay, an expected average of 2 weeks

SECONDARY OUTCOMES:
Mortality | Participants will be followed for the duration of intensive care unit stay, an expected average of 2 weeks
Days of mechanical ventilation | From date of randomization until the date of death or date of extubation, whichever comes first, an expected average of 2 weeks
Length of stay | From date of randomization until the date of death or date of discharge from the intensive care unit, an expected average of 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jesus J Martinez, MD, Study Chair — Sinaloa Pediatric Hospital
Locations (1):
- Sinaloa Pediatric Hospital, Culiacán, Sinaloa, Mexico